CLINICAL TRIAL: NCT03880630
Title: Inspiratory Muscle Activation Pattern Analysis in Assisting Precision in Inspiratory Muscle Training in Patients With Chronic Respiratory Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201812172RIND
Record Dates: First submitted 2019-03-14; First posted 2019-03-19 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2020-03

CONDITIONS: Chronic Respiratory Disease; Inspiratory Muscle Training; Sternocleidomastoid Muscle; Surface Electromyography

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chronic respiratory disease (Experimental): Patients with chronic respiratory disease with inspiratory muscle weakness will be recruited for the study
  Interventions: Other: Inspiratory muscle training

INTERVENTIONS:
Other: Inspiratory muscle training — Patients will perform 3 inspiratory loading tests (15%, 30%, and 50% of maximum inspiratory pressures) on 3 separate days with the sequence will be randomized. Patient will then be trained with individualized IMT program based on the results of 3 inspiratory loading tests.

SUMMARY:
Background & Objective: Inspiratory muscle training (IMT) is known to improve strength and endurance of inspiratory muscles. However, clinical beneficial effects of IMT for patients with chronic respiratory disease remain inconclusive.

The purposes of the study are to investigate in patients with chronic respiratory disease: (Year 1) main (diaphragm) and accessory inspiratory muscle (sternocleidomastoid muscle) activation pattern during various IMT loading using group-based trajectory modeling (GBTM); and (Year 2) effectiveness of individualized IMT program (based on results of Year 1) on clinical outcomes. Methods: (Year 1) Patients with chronic respiratory disease with inspiratory muscle weakness will be recruited for the study. Patients will perform 3 inspiratory loading tests (15%, 30%, and 50% of maximum inspiratory pressures) on 3 separate days with the sequence will be randomized. Surface electromyography (EMG) of diaphragm and sternocleidomastoid muscle will be used to use inspiratory muscle activation during various conditions. Other outcomes include maximum inspiratory pressure, and functional exercise capacity will be measured. Inspiratory muscle activation will be used for GBTM analysis. Patient will then be trained with individualized IMT program based on the GBTM analysis input form results of Year 1.

ELIGIBILITY:
Inclusion Criteria:

* age > 20 years old
* has been diagnosis of chronic obstructive pulmonary disease with stable clinical condition with no infection or acute exacerbation in the previous four weeks
* can cooperate with the measurements of this study

Exclusion Criteria:

* any clinical diagnosis that will influence the measurement, including any history of
* neuromyopathy
* angina, acute myocardial infarction in the previous one month
* pregnancy
* participated in inspiratory muscle training program in the previous three months
* any psychiatric or cognitive disorders, for example: Mini-Mental State Examination (MMSE) < 24, that will disturb the communication and cooperation of the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-10-06 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Diaphragm and Sternocleidomastoid muscle activation | through the completion of the inspiratory loading tests condition; it would take about 3 minutes
  Root mean square values during different conditions
The mean median frequency of diaphragm and sternocleidomastoid muscle | In five minute after the completion of the loaded inspiratory muscle test condition
  The power spectrum is divided into two equal areas of the frequency value by median frequency to exam muscle fatigability
Pulmonary function | About five minutes to complete
  Forced expiratory volume in one second, forced vital capacity, residual volume, total lung capacity
Maximal inspiratory pressure test | About three minutes to complete
  Maximal inspiratory pressure
Functional exercise capacity using the six-minute walk test | The six-minute walk test needs six minute to complete the test
  The six-minute walk test is commonly performed to evaluate functional exercise capacity. The six-minute walk test was performed according to the guidelines, and the distance walked in the test presented as functional exercise capacity
Heart rate | The six-minute walk test needs six minute to complete the test
  Heart rate is measured at rest, during six-minute walk test
Blood pressure | Before and immediately after the six-minute walk test;it takes less than one minute to measure blood pressure
  systolic and diastolic pressure are measured at rest, after six-minute walk test
Perceived dyspnea | It takes less than one minute to evaluate perceived dyspnea
  Rating of perceived dyspnea is measured by using Borg scale at rest, during six-minute walk test, inspiratory loading tests. The most widely used tool is the "Borg scale", with rating ranges from 0 (nothing at all) to 10 (extremely dyspnea).
Oxygen saturation | The six-minute walk test needs six minute to complete the test; through the completion of the inspiratory loading tests condition; it would take about 3 minutes
  Oxygen saturation is continuously monitored by pulse oximetry throughout six-minute walk test, inspiratory loading tests

CONTACTS AND LOCATIONS:
Overall Officials: Li-Ying Wang, Phd, Study Chair — National Taiwan University
Locations (1):
- School & Graduate Institute of Physical Therapy, College of Medicine, NTU, Taipei, Taiwan